CLINICAL TRIAL: NCT00660010
Title: Study of Lupron Depot In The Treatment of Central Precocious Puberty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Kristof Chwalisz, MD, PhD Therapeutic Area Head, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M90-516
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Results first posted 2010-07-20 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Puberty, Precocious
Keywords: CPP; central precocious puberty; pediatrics; suppression of LH; Lupron; leuprolide acetate; depot formulation; GnRHa; GnRH agonist; GNRH analog; LH; Tanner staging
MeSH Terms: conditions — Puberty, Precocious | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Lupron (leuprolide acetate)

INTERVENTIONS:
Drug: Lupron (leuprolide acetate) — Leuprolide acetate was administered monthly by intramuscular injection starting at 300 mcg/kg with adjustments of 3.75 mg upward, at subsequent clinic visits based on physical and laboratory parameters. Dosing continued until NDA was approved, or until subject no longer required leuprolide acetate to treat CPP.
  Other Names: Lupron

SUMMARY:
The purpose of this study is to determine if Lupron (leuprolide acetate) is safe and effective in treating children with Central Precocious Puberty (CPP), and to assess long term effects of leuprolide acetate treatment after therapy is discontinued.

DETAILED DESCRIPTION:
This study includes a Prestudy Period; a treatment period where subjects will receive treatment every 4 weeks until the initiation of puberty (age 12 for males and age 11 for females); a follow-up period where subjects will be observed every 6 months until physical and laboratory observations are at pubertal levels, then every 12 months for 5 years; lastly a final follow-up questionnaire is given to all subjects when they are at least 18 years old.

At the treatment visits, efficacy assessments are Tanner staging (suppression of breast development in females and genital development in males), gonadotropins (LH and FSH), sex steroids (estradiol in females and testosterone in males), ratio of bone age to chronological age, adult height compared to a standard population and predicted mature height, and age and time to regular menses in females. This protocol will also capture data from the final questionnaire about female reproductive status at adulthood including the presence of regular menses and number of pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of isosexual central precocious puberty with onset of Tanner scores of Stage II for breast or pubic hair earlier than age 8.0 years in girls or Stage II for pubic hair or genitalia earlier than 9.0 years in boys.
* Confirmation of diagnosis by a pubertal response to a gonadotropin-releasing hormone (GnRH) stimulation test (LH > 10 U/L at baseline).
* Chronological age less than 9.0 years in girls or less than 10.0 years in boys at time of first dosing.
* Bone age advanced at least 1 year beyond the chronological age at entry into the study.
* The condition may be idiopathic or secondary to another lesion. If secondary, therapy of the primary condition will have been undertaken and stabilized.
* No evidence of abnormal pituitary, adrenal, thyroid and gonadal function except for premature secretion of gonadotropins.

Exclusion Criteria:

* Irradiation to the central nervous system.
* Prior therapy with medroxyprogesterone acetate and/or with any GnRH analog (including prior treatment with daily subcutaneous and depot formulations of leuprolide acetate).

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 1991-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristof Chwalisz, MD, Study Director — Abbott
Locations (9):
- United States (9):
  - Site Reference ID/Investigator# 46673, Phoenix, Arizona
  - Site Reference ID/Investigator# 46671, San Francisco, California
  - Site Reference ID/Investigator# 14921, Stanford, California
  - Site Reference ID/Investigator# 14343, Aurora, Colorado
  - Site Reference ID/Investigator# 14341, St. Petersburg, Florida
  - Site Reference ID/Investigator# 14342, Indianapolis, Indiana
  - Site Reference ID/Investigator# 46672, Baltimore, Maryland
  - Site Reference ID/Investigator# 46668, Springfield, Massachusetts
  - Site Reference ID/Investigator# 14344, Hershey, Pennsylvania

REFERENCES:
- [Derived] Lee PA, Neely EK, Fuqua J, Yang D, Larsen LM, Mattia-Goldberg C, Chwalisz K. Efficacy of Leuprolide Acetate 1-Month Depot for Central Precocious Puberty (CPP): Growth Outcomes During a Prospective, Longitudinal Study. Int J Pediatr Endocrinol. 2011;2011(1):7. doi: 10.1186/1687-9856-2011-7. Epub 2011 Jul 12. PMID 21860633

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included 1 treatment group and subjects were assigned the initial dosage depending on their weight. The minimum starting dose was 7.5 mg every 28 days. Study drug was discontinued either when puberty occurred at 12 years +- 6 months for males and 11 years +- 6 months for females or at the discretion of the investigator.
Groups:
- Leuprolide Acetate 1 Month Depot: Leuprolide acetate dosing was initiated at 300 mcg/kg (minimum dose 7.5 mg) administered intramuscularly (IM) every 28 days. Incremental adjustments to dosing at 3.75 mg increments were made at each visit.
Period: Overall Study
Arm/Group | Leuprolide Acetate 1 Month Depot
Started | 55
Completed | 46
Not Completed | 9
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 1
Not completed — Noncompliance with visit schedule | 3

BASELINE CHARACTERISTICS:
Arm/Group | Leuprolide Acetate 1 Month Depot
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 55
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 6.9 (1.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 6
Region of Enrollment [Number; unit: subjects]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects (n/N) With Suppression of Clinical Sexual Characteristics According to Tanner Staging (Breast Development in Females)
Description: Suppression of clinical sexual characteristics was defined as regression (improvement) or no progression of breast development in females. Tanner staging is a scale of physical development that defines primary and secondary sex characteristics including size of breasts. The final visit occurred at a mean age +/- SD of 11.05 +/- 1.14 years (range, 6.96 to 12.95 years).
Time Frame: Week 4, Week 48 (Year 1), yearly for 5 years (Week 240), and Final Visit
Population: The intent-to-treat (ITT) population and safety analysis set were identical for the treatment period. The starting population comprised 49 females (breast development suppression). Study drug was discontinued at the initiation of puberty.
Measure: Number; unit: Percentage of subjects
Arm/Group | Leuprolide Acetate 1 Month Depot
Number analyzed (Participants) | 49
Percentage of subjects
  Breast development suppression - Week 4 N=44 | 81.8
  Breast development suppression-Week 48 N=47 | 80.9 [66.7 to 90.9]
  Breast development suppression -Week 96 N=41 | 87.8 [73.8 to 95.9]
  Breast development suppression-Week 144 N=29 | 82.8 [64.2 to 94.2]
  Breast development suppression - Week 192 N=18 | 66.7 [41.0 to 86.7]
  Breast development suppression -Week 240 N=13 | 76.9 [46.2 to 95.0]
  Breast development suppression-Final Visit N=48 | 77.1

2. Secondary Outcome: Mean Peak Stimulated Luteinizing Hormone (LH) and Follicle Stimulating Hormone (FSH) Concentrations
Description: Mean peak stimulated visit LH and FSH concentrations were assessed according to the DELFIA (registered trademark) assay. The final visit for measurement of both hormone concentrations occurred at a mean age +/- SD of 11.13 +/- 1.23 (range, 6.73 to 14.07) years.
Time Frame: Baseline, Weeks 4, 12, 24, 48 (Year 1), yearly for 5 years (Week 240), and Final Visit
Population: The intent-to-treat (ITT) population and safety analysis set were identical for the treatment period. The starting population comprised 49 females and 6 males. Study drug was discontinued at the initiation of puberty.
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Leuprolide Acetate 1 Month Depot
Number analyzed (Participants) | 55
mIU/mL
  Peak stimulated LH at Baseline N=55 | 35.0 (21.32)
  Peak stimulated LH at Week 4 N = 55 | 0.8 (0.57)
  Peak stimulated LH at Week 12 N = 54 | 1.1 (1.77)
  Peak stimulated LH at Week 24 N = 53 | 0.8 (0.79)
  Peak stimulated LH at Week 48 N = 54 | 0.6 (0.47)
  Peak stimulated LH at Week 96 N = 46 | 0.4 (0.33)
  Peak stimulated LH at Week 144 N = 36 | 0.4 (0.24)
  Peak stimulated LH at Week 192 N = 20 | 0.4 (0.25)
  Peak stimulated LH at Week 240 N = 17 | 0.4 (0.62)
  Peak stimulated LH at Final Visit N = 55 | 0.8 (3.29)
  Peak stimulated FSH at Baseline N=55 | 13.3 (5.58)
  Peak stimulated FSH at Week 4 N = 55 | 0.9 (0.44)
  Peak stimulated FSH at Week 12 N = 54 | 1.1 (0.61)
  Peak stimulated FSH at Week 24 N = 53 | 1.2 (0.84)
  Peak stimulated FSH at Week 48 N = 54 | 1.2 (0.58)
  Peak stimulated FSH at Week 96 N = 46 | 1.4 (0.79)
  Peak stimulated FSH at Week 144 N = 36 | 1.4 (0.73)
  Peak stimulated FSH at Week 192 N = 20 | 1.3 (0.76)
  Peak stimulated FSH at Week 240 N = 17 | 1.4 (0.67)
  Peak stimulated FSH at Final Visit N = 55 | 1.7 (1.73)

3. Secondary Outcome: Mean Stimulated Estradiol Concentrations in Females
Description: Mean estradiol concentrations were assessed according to the DELFIA (registered trademark) assay. The lower limit of quantitation for estradiol is 5 pg/mL and measurements below this limit are given a value of 5 pg/mL. The final visit for measurement estradiol concentrations occurred at a mean age +/- SD of 10.93 +/- 1.27 (range, 5.59 to 13.24) years.
Time Frame: Baseline, Weeks 4, 12, 24, 48 (Year 1), yearly for 5 years (Week 240), and Final Visit
Population: All females in the intent-to-treat (ITT) population and safety analysis set were identical for the treatment period. Study drug was discontinued at the initiation of puberty.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Leuprolide Acetate 1 Month Depot
Number analyzed (Participants) | 49
pg/mL
  Mean stimulated estradiol at baseline N=49 | 15.3 (18.73)
  Mean stimulated estradiol at Week 4 N=48 | 5.0 (0.00)
  Mean stimulated estradiol at Week 12 N=47 | 6.0 (6.56)
  Mean stimulated estradiol at Week 24 N=47 | 5.0 (0.00)
  Mean stimulated estradiol at Week 48 N=47 | 5.0 (0.00)
  Mean stimulated estradiol at Week 96 N=39 | 5.0 (0.00)
  Mean stimulated estradiol at Week 144 N=31 | 5.0 (0.00)
  Mean stimulated estradiol at Week 192 N=15 | 5.0 (0.00)
  Mean stimulated estradiol at Week 240 N=13 | 5.0 (0.00)
  Mean stimulated estradiol at Final Visit N=49 | 5.0 (0.14)

4. Secondary Outcome: Mean Stimulated Testosterone Concentrations in Males
Description: Mean stimulated testosterone concentrations were assessed according to the DELFIA (registered trademark) assay. The final visit for measurement of testosterone occurred at a mean age +/- SD of 12.34 +/- 1.16 (range, 11.14 to 14.07) years.
Time Frame: Baseline, Weeks 4, 12, 24, 48 (Year 1), yearly for 5 years (Week 240), and Final Visit
Population: All males in the intent-to-treat (ITT) population and safety analysis set were identical for the treatment period. Study drug was discontinued at the initiation of puberty.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Leuprolide Acetate 1 Month Depot
Number analyzed (Participants) | 6
ng/dL
  Mean stimulated testosterone at baseline N=6 | 347.7 (121.86)
  Mean stimulated testosterone at Week 4 N=6 | 18.0 (12.39)
  Mean stimulated testosterone at Week 12 N=6 | 14.2 (7.05)
  Mean stimulated testosterone at Week 24 N=6 | 13.8 (6.15)
  Mean stimulated testosterone at Week 48 N=6 | 17.3 (11.64)
  Mean stimulated testosterone at Week 96 N=6 | 24.8 (19.92)
  Mean stimulated testosterone at Week 144 N=5 | 21.6 (19.50)
  Mean stimulated testosterone at Week 192 N=4 | 24.0 (17.19)
  Mean stimulated testosterone at Week 240 N=3 | 25.3 (24.01)
  Mean stimulated testosterone at Final Visit N=6 | 24.2 (17.16)

5. Secondary Outcome: Mean Ratio of Bone Age to Chronological Age
Description: Bone age was determined by radiography of the wrist according to the Fels Method. The mean ratio of bone age to chronological age provides information about the slowing of bone age progression. A score = 1 indicates that bone age is equal to chronological age.
Time Frame: Week 24 and Week 48 (Year 1), yearly for 5 years (Week 240), and Final Visit
Population: The intent-to-treat (ITT) population and safety analysis set were identical for the treatment period. Study drug was discontinued at the initiation of puberty.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Leuprolide Acetate 1 Month Depot
Number analyzed (Participants) | 53
ratio
  Ratio at Baseline N=53 | 1.5 (0.30)
  Ratio at Week 24 N=53 | 1.5 (0.25)
  Ratio at Week 48 N=51 | 1.4 (0.18)
  Ratio at Week 96 N=44 | 1.3 (0.15)
  Ratio at Week 144 N=31 | 1.2 (0.12)
  Ratio at Week 192 N=26 | 1.2 (0.11)
  Ratio at Week 240 N=16 | 1.2 (0.10)
  Ratio at Final Visit N=53 | 1.2 (0.11)

6. Other Pre Specified Outcome: Posttreatment Height (ht.) Compared to Standard Population and as Predicted From Ht. at Baseline (BL)
Description: Height was measured by stadiometer and was standardized for age according to standard growth charts. A standardized score of 0 indicated a mean ht. equivalent to mean of a standard population from 2000 CDC standardized ht. charts. Height gain was calculated as ht. - predicted ht. from the Bayley-Pinneau method on the basis of bone age at baseline. Final adult ht. was determined by measurement at final adult ht., if available, or by ht. collected during the follow-up period associated with a growth velocity <1 cm/year or a bone age >14 yrs in females or >15 yrs in males.
Time Frame: Final ht. (measured or provided for final questionnaire in subjects >= 18 years of age) or near final adult ht. (<1 cm/year or bone age > 14 years for females or > 15 years for males)
Population: For the follow-up posttreatment period, the ITT population=40 subjects and the safety population=55 subjects who received at least 1 injection of study drug during the treatment period. Study drug was discontinued at the initiation of puberty. The mean age of subjects at final questionnaire completion was 24.76 years with a range of 18.87 to 26.66.
Measure: Mean (Standard Error); unit: cm
Arm/Group | Leuprolide Acetate 1 Month Depot
Number analyzed (Participants) | 40
cm
  Near final adult ht. standardized score N=33 | -0.2 (1.20)
  Near final ht.gain from predicted ht. at BL N=29 | 3.2 (5.37)
  Final adult ht.standardized score N=19 | 0.0 (1.13)
  Final adult ht.gain from predicted ht. at BL N=17 | 3.9 (5.05)

7. Other Pre Specified Outcome: Mean Time to or Mean Age at Regular Menses in Females After Treatment
Description: Regular menses was defined as 3 or more consecutive days of menstrual-like bleeding and was defined by the investigator's clinical judgment.
Time Frame: Posttreatment during the follow-up period (subjects observed every 6 months until physical and laboratory observations are at pubertal levels)
Population: During the posttreatment period, data were obtained from 32 female subjects. Twenty-seven subjects reported the start of menses, but only 26 subjects reported a menses start date.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Leuprolide Acetate 1 Month Depot
Number analyzed (Participants) | 26
years
  Time to regular menses | 1.5 (0.53)
  Age at regular menses | 12.9 (0.89)

8. Other Pre Specified Outcome: Number of Female Subjects Who Reported Regular Menses at Adulthood
Description: Subjects were required to complete final adult questionnaire to provide information on adult reproductive function. Regular menses was defined as 3 or more consecutive days of menstrual-like bleeding.
Time Frame: Posttreatment data were collected from the final adult questionnaire (subjects >= 18 years of age)
Population: A long-term follow-up questionnaire was sent to all subjects who completed at least 1 visit in the posttreatment follow-up period or who discontinued treatment because they entered puberty naturally at the appropriate age. Twenty female subjects (mean age 24.76 years, range 18.87 to 26.66 years) and 0 male subjects completed the questionnaire.
Measure: Number; unit: Subjects
Arm/Group | Leuprolide Acetate 1 Month Depot
Number analyzed (Participants) | 20
Subjects
  No. of subjects with regular menses as adults | 16
  No. of subjects without regular menses as adults | 4

9. Other Pre Specified Outcome: Number of Subjects Who Reported Pregnancies at Final Questionnaire
Description: The final questionnaire was completed by 20 females who were at least 18 years of age. The subjects reported on total number of pregnancies resulting in live births or number of miscarriages (spontaneous or elective) and whether the subject was currently pregnant.
Time Frame: Posttreatment data were collected from the final adult questionnaire (subjects >= 18 years of age)
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | Leuprolide Acetate 1 Month Depot
Number analyzed (Participants) | 20
Subjects
  Number of subjects who reported being pregnant | 7
  Number of subjects who were currently pregnant | 1

10. Other Pre Specified Outcome: Number of Pregnancies Reported by Subjects at Final Questionnaire
Description: The final questionnaire was completed by 20 female subjects who were at least 18 years of age. The total number of pregnancies were reported.
Time Frame: Posttreatment data were collected from the final adult questionnaire (subjects >= 18 years of age)
Population: as for outcome 8
Measure: Number; unit: Pregnancies
Arm/Group | Leuprolide Acetate 1 Month Depot
Number analyzed (Participants) | 20
Pregnancies
  Number of pregnancies | 12
  Number of live births | 6
  Number of miscarriages | 5

11. Primary Outcome: Percentage of Subjects (n/N) With Suppression of Clinical Sexual Characteristics According to Tanner Staging (Genital Development in Males)
Description: Suppression of clinical sexual characteristics was defined as regression (improvement) or no progression of genital development in males. Tanner staging is a scale of physical development that defines primary and secondary sex characteristics including size of genitals. The final visit occurred at a mean age +/- SD of 12.35 +/-1.35 years (range, 10.71 to 14.07 years).
Time Frame: Week 4, Week 48 (Year 1), yearly for 5 years (Week 240), and Final Visit
Population: The intent-to-treat (ITT) population and safety analysis set were identical for the treatment period. The starting population comprised 6 males (genital development suppression). Study drug was discontinued at the initiation of puberty.
Measure: Number; unit: Percentage of subjects
Arm/Group | Leuprolide Acetate 1 Month Depot
Number analyzed (Participants) | 6
Percentage of subjects
  Genital development suppression - Week 4 N=5 | 80.0
  Genital development suppression - Week 48 N=6 | 83.3
  Genital development suppression - Week 96 N=6 | 83.3
  Genital development suppression - Week 144 N=4 | 75.0
  Genital development suppression - Week 192 N=4 | 75.0
  Genital development suppression - Week 240 N=3 | 66.7
  Genital development suppression - Final Visit N=6 | 83.3

ADVERSE EVENTS:
Time Frame: Each investigator monitored each subject for clinical and laboratory evidence of adverse events at Weeks 4, 8, 12, 24, 36, 48, and then every 6 months until the study drug was discontinued.
Description: Adverse events were reported from onset after the first injection of study drug through 30 days after treatment was completed. Treatment completion was defined as 28 days after the final study drug injection. The posttreatment follow-up period did not require the reporting of adverse events.
Arm/Group | Leuprolide Acetate 1 Month Depot
Serious Adverse Events (participants affected / at risk) | 7/55
Other Adverse Events (participants affected / at risk) | 52/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprolide Acetate 1 Month Depot (N=55)
Aggravation reaction (General disorders) | 1 — COSTART body system is body as a whole
Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — COSTART body system is body as a whole
Infection (Infections and infestations) | 1 — COSTART body system is body as a whole
Heart arrest (Cardiac disorders) | 1 — COSTART body system is cardiovascular system
Bone Disorder (Musculoskeletal and connective tissue disorders) | 1 — COSTART body system is musculoskeletal system
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 — COSTART body system is musculoskeletal system
Personality disorder (Psychiatric disorders) | 1 — COSTART body system is nervous system
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 — COSTART body system is respiratory system
Pneumonia (Infections and infestations) | 1 — COSTART body system is respiratory system
Repair of ventriculoperitoneal shunt (Surgical and medical procedures) | 1 — COSTART body system was not classified since it was a surgical repair.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprolide Acetate 1 Month Depot (N=55)
Abdominal pain (Gastrointestinal disorders) | 16 — COSTART body system is body as a whole
Accidental injury (Injury, poisoning and procedural complications) | 16 — COSTART body system is body as a whole
Allergic reaction (Immune system disorders) | 6 — COSTART body system is body as a whole
Asthenia (General disorders) | 6 — COSTART body system is body as a whole
Body odor (Skin and subcutaneous tissue disorders) | 3 — COSTART body system is body as a whole
Fever (General disorders) | 14 — COSTART body system is body as a whole
Flu syndrome (Infections and infestations) | 19 — COSTART body system is body as a whole
Headache (Nervous system disorders) | 25 — COSTART body system is body as a whole
Infection (Infections and infestations) | 13 — COSTART body system is body as a whole
Injection site pain (General disorders) | 8 — COSTART body system is body as a whole
Injection site reaction (General disorders) | 3 — COSTART body system is body as a whole
Pain (General disorders) | 12 — COSTART body system is body as a whole
Reaction unevaluable (General disorders) | 5 — COSTART body system is body as a whole
Vasodilatation (Vascular disorders) | 6 — COSTART body system is cardiovascular system
Diarrhea (Gastrointestinal disorders) | 9 — COSTART body system is digestive system
Dyspepsia (Gastrointestinal disorders) | 5 — COSTART body system is digestive system
Increased appetite (Metabolism and nutrition disorders) | 5 — COSTART body system is digestive system
Nausea (Gastrointestinal disorders) | 7 — COSTART body system is digestive system
Vomiting (Gastrointestinal disorders) | 13 — COSTART body system is digestive system
Lymphadenopathy (Blood and lymphatic system disorders) | 3 — COSTART body system is hemic and lymphatic system
Edema (General disorders) | 4 — COSTART body system is metabolic and nutritional disorders
Growth retarded (Musculoskeletal and connective tissue disorders) | 6 — COSTART body system is metabolic and nutritional disorders
Weight gain (Investigations) | 9 — COSTART body system is metabolic and nutritional disorders
Weight loss (Investigations) | 3 — COSTART body system is metabolic and nutritional disorders
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 — COSTART body system is musculoskeletal system
Myalgia (Musculoskeletal and connective tissue disorders) | 4 — COSTART body system is musculoskeletal system
Pathological fracture (Musculoskeletal and connective tissue disorders) | 4 — COSTART body system is musculoskeletal system
Depression (Psychiatric disorders) | 3 — COSTART body system is nervous system
Dizziness (Nervous system disorders) | 4 — COSTART body system is nervous system
Emotional Lability (Psychiatric disorders) | 15 — COSTART body system is nervous system
Nervousness (Psychiatric disorders) | 4 — COSTART body system is nervous system
Cough increased (Respiratory, thoracic and mediastinal disorders) | 17 — COSTART body system is respiratory system
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 — COSTART body system is respiratory system
Pharyngitis (Infections and infestations) | 29 — COSTART body system is respiratory system
Rhinitis (Infections and infestations) | 14 — COSTART body system is respiratory system
Sinusitis (Infections and infestations) | 11 — COSTART body system is respiratory system
Acne (Skin and subcutaneous tissue disorders) | 15 — COSTART body system is skin and appendages
Herpes zoster (Infections and infestations) | 8 — COSTART body system is skin and appendages
Hirsutism (Skin and subcutaneous tissue disorders) | 3 — COSTART body system is skin and appendages
Pruritus (Skin and subcutaneous tissue disorders) | 3 — COSTART body system is skin and appendages
Rash (Skin and subcutaneous tissue disorders) | 18 — COSTART body system is skin and appendages
Skin disorder (Skin and subcutaneous tissue disorders) | 6 — COSTART body system is skin and appendages
Urticaria (Skin and subcutaneous tissue disorders) | 4 — COSTART body system is skin and appendages
Ear pain (Ear and labyrinth disorders) | 4 — COSTART body system is special senses
Eye disorder (Eye disorders) | 3 — COSTART body system is special senses
Otitis media (Infections and infestations) | 15 — COSTART body system is special senses
Leukorrhea (Reproductive system and breast disorders) | 4 — COSTART body system is urogenital system
Menstrual disorder (Reproductive system and breast disorders) | 3 — COSTART body system is urogenital system
Urinary tract infection (Infections and infestations) | 4 — COSTART body system is urogenital system
Vaginitis (Infections and infestations) | 11 — COSTART body system is urogenital system

LIMITATIONS AND CAVEATS:
Study drug was discontinued usually at the initiation of puberty (12 years for males and 11 years for females) with the concurrence of the investigator, or at the discretion of the investigator. Adverse events are coded with the COSTART dictionary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.